CLINICAL TRIAL: NCT02959255
Title: A Greek, Single Center, Randomized, Double Blind Controlled Clinical Study Comparing the 10-day Versus the 14-day Concomitant Proton Pump Inhibitor [PPI] + Amoxicillin + Metronidazole + Clarithromycin (PAMC) Therapeutic Scheme as First-line Treatment Strategy for the Eradication of H. Pylori Infection
Brief Title: 10-day Versus 14-day Concomitant PAMC as First-line Treatment Strategy for the Eradication of H. Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS-EL-ESO-2016
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10-day concomitant PAMC (Active Comparator): 40mg esomeprazole twice daily, 500mg clarithromycin twice daily, 1gr amoxicillin twice daily, and 500mg metronidazole twice daily for 10 days
  Interventions: Drug: Esomeprazole
- 14-day concomitant PAMC (Active Comparator): (40mg esomeprazole twice daily, 500mg clarithromycin twice daily, 1gr amoxicillin twice daily, and 500mg metronidazole twice daily for 14 days.
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — dosage difference

SUMMARY:
Helicobacter pylori (H. pylori) infection is highly associated with gastrointestinal disorders, including peptic ulcer disease, gastric cancer, and gastric mucosa associated lymphoid tissue lymphoma.1 In 1994, H. pylori was classified as a group carcinogen by the International Agency for Research on Cancer. Since then, many consensus conferences and clinical guidelines worldwide have been established for the treatment of H. pylori infection.

Despite H. pylori infecting an estimated 50% of the global population,there is no universally effective regimen in everyday clinical practice. The current European Helicobacter Study Group Guidelines for the first line empirical treatment of the H. pylori infection propose a variety of treatment strategies, as optimal treatment of H. pylori infection requires careful attention to local antibiotic resistance and eradication patterns. Most recently, the Toronto Consensus for the Treatment of Helicobacter pylori Infection in Adults strongly recommended that all H. pylori eradication regimens now be given for 14 days. Recommended first-line strategies include concomitant nonbismuth quadruple therapy (proton pump inhibitor [PPI] + amoxicillin + metronidazole + clarithromycin [PAMC]) and traditional bismuth quadruple therapy (PPI + bismuth + metronidazole + tetracycline [PBMT]).The aforementioned statement by an international working group of specialists chosen by the Canadian Association of Gastroenterology is of the outmost importance, especially in countries with increased antibiotic resistance, like Greece, with resistance rates >20% to clarithromycin and >40% to metronidazole.

DETAILED DESCRIPTION:
In Greece, while the efficacy of the 10-day concomitant PAMC scheme has been recently established,to our knowledge no head-to-head comparison evaluating treatment time (10 versus 14 days) of the same therapeutic regimen has been tried out. We decided to conduct a randomized double blind controlled clinical study comparing the 10-day versus the 14-day concomitant PAMC therapeutic scheme as first-line treatment strategy for the eradication of H. pylori infection, in a country of increased dual resistance to clarithromycin and metronidazole (where bismuth is unavailable). The primary end point of our study will be treatment efficacy (primary and secondary antibiotic resistance), while secondary end points will be patient compliance and safety.

This open labeled prospective randomized trial will be held at the Army Share Fund Hospital (NIMTS), in Athens, Greece, and will be conducted by the Hospital's Department of Gastroenterology. Written informed consent will obtained from all participants before enrollment. The study must be approved before hand by the Institutional Review Board of Hospital.

Interventions A physician will be recruited so as to obtain the patients' demographic data and medical history. Using sealed envelopes, eligible patients will be randomized in two groups, with a research assistant assigning the therapies according to the treatment allocations kept in the envelopes. In the first group, patients will be assigned to a 10-day concomitant PAMC therapy (40mg esomeprazole twice daily, 500mg clarithromycin twice daily, 1gr amoxicillin twice daily, and 500mg metronidazole twice daily). In the second group, patients will be assigned to the same concomitant PAMC therapy for 14days. Each envelope will contain precise written instructions regarding the treatment schedule, dosing, and time of medication ingestion, while further instructions will be available, if needed, via the telephone.

Follow-up and outcome To confirm compliance, all patients will be asked to bring their remaining medication 5 days after the end of the treatment where we will count the rest of their pills. Patients with a compliance <80% will be excluded from the study per protocol (PP) analysis. Patients will also be interviewed for reasons responsible for missing any doses of the regimens, as well as for the occurrence of any new or worsened medical conditions that led them to seek medical attention. Adverse events will be classified as minor or major, with the later leading to discontinuation of the treatment.

Four weeks after the treatment period (with no administration of PPIs or any antibiotics), we will confirm H. pylori eradication using C13-UBT by a staff member who will be blind to the eradication arm of each patient. In case of treatment failure, a repeated endoscopy will be performed with biopsy specimens being taken (two from the antrum and two from the body of the stomach). Biopsy specimens will be cultured and antibiotic susceptibility will be determined for amoxicillin, tetracycline, clarithromycin, metronidazole, and levofloxacin with the aid of the agar dilution test, according to the standard European protocol.14,15 The microbiologist who will be performing the agar dilution test will be blinded to the treatment. If first-line eradication therapy fails, second-line therapy will be administered, according to antibiotic susceptibility.

Statistical analysis In this study, a clinically significant difference for eradication between the two groups will be 15%. In order to achieve 80% power for detecting this difference, along with an alpha level of 0.05 and an allocation ratio of 1:1, we calculated a needed sample of 364 patients. Since this is a convenient clinical sample, the study will be terminated either by reaching this number of patients or by the study's timeline limitation. Baseline characteristics will be compared and the difference of the observed eradication rates between the study groups will be assessed. The results of this study will be analyzed in an intention to treat (ITT) and a PP population. The ITT analysis will include all randomized patients who will have taken at least one dose of the study medication (regardless of compliance). The patients whose infection statuses will be unknown following treatment will be considered treatment failures for the purposes of the ITT analysis. The PP analysis will include patients with at least 80% compliance (excluding the patients with unknown H. pylori status following therapy and those with major protocol violations).

ELIGIBILITY:
Inclusion Criteria:

* age >18 or <80 years
* consecutive newly diagnosed H. pylori-infected patients
* endoscopically proven peptic ulcer disease or non-ulcer dyspepsia
* H. pylori infection will be established by at least one positive test among C13-urea breath test (UBT), rapid urease test, and gastric histology.
* patients who have signed the Informed Consent
* patients who will be compliant to study procedures

Exclusion Criteria:

* age <18 or >80 years.
* previous H. pylori eradication therapy
* known allergic history to any of the medications used in our study
* pregnancy or lactation
* ingestion of antibiotics within the prior 4 weeks
* patients with previous gastric surgery
* the coexistence of serious concomitant illness which would not allow patients' compliance (i.e., malignant neoplasms)
* addiction to alcohol or illicit and recreational drugs
* patients who have not signed Informed Consent
* patients who will not comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Helicobacter Pylori eradication | 10 days - 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Army Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papastergiou V, Georgopoulos SD, Karatapanis S. Treatment of Helicobacter pylori infection: Past, present and future. World J Gastrointest Pathophysiol. 2014 Nov 15;5(4):392-9. doi: 10.4291/wjgp.v5.i4.392. PMID 25400982
- [Background] Schistosomes, liver flukes and Helicobacter pylori. IARC Monogr Eval Carcinog Risks Hum. 1994;61:1-241. No abstract available. PMID 7715068
- [Background] Infection with Helicobacter pylori. IARC Monogr Eval Carcinog Risks Hum. 1994;61:177-240. No abstract available. PMID 7715070
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] World Gastroenterology Organisation. World Gastroenterology Organisation Global Guideline: Helicobacter pylori in developing countries. J Clin Gastroenterol. 2011 May-Jun;45(5):383-8. doi: 10.1097/MCG.0b013e31820fb8f6. No abstract available. PMID 21415768
- [Background] Fock KM, Katelaris P, Sugano K, Ang TL, Hunt R, Talley NJ, Lam SK, Xiao SD, Tan HJ, Wu CY, Jung HC, Hoang BH, Kachintorn U, Goh KL, Chiba T, Rani AA; Second Asia-Pacific Conference. Second Asia-Pacific Consensus Guidelines for Helicobacter pylori infection. J Gastroenterol Hepatol. 2009 Oct;24(10):1587-600. doi: 10.1111/j.1440-1746.2009.05982.x. PMID 19788600
- [Background] Chey WD, Wong BC; Practice Parameters Committee of the American College of Gastroenterology. American College of Gastroenterology guideline on the management of Helicobacter pylori infection. Am J Gastroenterol. 2007 Aug;102(8):1808-25. doi: 10.1111/j.1572-0241.2007.01393.x. Epub 2007 Jun 29. PMID 17608775
- [Background] Watari J, Chen N, Amenta PS, Fukui H, Oshima T, Tomita T, Miwa H, Lim KJ, Das KM. Helicobacter pylori associated chronic gastritis, clinical syndromes, precancerous lesions, and pathogenesis of gastric cancer development. World J Gastroenterol. 2014 May 14;20(18):5461-73. doi: 10.3748/wjg.v20.i18.5461. PMID 24833876
- [Background] De Francesco V, Giorgio F, Hassan C, Manes G, Vannella L, Panella C, Ierardi E, Zullo A. Worldwide H. pylori antibiotic resistance: a systematic review. J Gastrointestin Liver Dis. 2010 Dec;19(4):409-14. PMID 21188333
- [Background] Papastergiou V, Georgopoulos SD, Karatapanis S. Treatment of Helicobacter pylori infection: meeting the challenge of antimicrobial resistance. World J Gastroenterol. 2014 Aug 7;20(29):9898-911. doi: 10.3748/wjg.v20.i29.9898. PMID 25110420
- [Background] Fallone CA, Chiba N, van Zanten SV, Fischbach L, Gisbert JP, Hunt RH, Jones NL, Render C, Leontiadis GI, Moayyedi P, Marshall JK. The Toronto Consensus for the Treatment of Helicobacter pylori Infection in Adults. Gastroenterology. 2016 Jul;151(1):51-69.e14. doi: 10.1053/j.gastro.2016.04.006. Epub 2016 Apr 19. PMID 27102658
- [Background] Karamanolis GP, Daikos GL, Xouris D, Goukos D, Delladetsima I, Ladas SD. The evolution of Helicobacter pylori antibiotics resistance over 10 years in Greece. Digestion. 2014;90(4):229-31. doi: 10.1159/000369898. Epub 2014 Dec 12. PMID 25531953
- [Background] Megraud F, Coenen S, Versporten A, Kist M, Lopez-Brea M, Hirschl AM, Andersen LP, Goossens H, Glupczynski Y; Study Group participants. Helicobacter pylori resistance to antibiotics in Europe and its relationship to antibiotic consumption. Gut. 2013 Jan;62(1):34-42. doi: 10.1136/gutjnl-2012-302254. Epub 2012 May 12. PMID 22580412
- [Background] Apostolopoulos P, Koumoutsos I, Ekmektzoglou K, Dogantzis P, Vlachou E, Kalantzis C, Tsibouris P, Alexandrakis G. Concomitant versus sequential therapy for the treatment of Helicobacter pylori infection: a Greek randomized prospective study. Scand J Gastroenterol. 2016;51(2):145-51. doi: 10.3109/00365521.2015.1079646. Epub 2015 Oct 5. PMID 26435055
- [Background] Zullo A, Vaira D, Vakil N, Hassan C, Gatta L, Ricci C, De Francesco V, Menegatti M, Tampieri A, Perna F, Rinaldi V, Perri F, Papadia C, Fornari F, Pilati S, Mete LS, Merla A, Poti R, Marinone G, Savioli A, Campo SM, Faleo D, Ierardi E, Miglioli M, Morini S. High eradication rates of Helicobacter pylori with a new sequential treatment. Aliment Pharmacol Ther. 2003 Mar 1;17(5):719-26. doi: 10.1046/j.1365-2036.2003.01461.x. PMID 12641522
- [Background] Boyanova L, Mentis A, Gubina M, Rozynek E, Gosciniak G, Kalenic S, Goral V, Kupcinskas L, Kantarceken B, Aydin A, Archimandritis A, Dzierzanowska D, Vcev A, Ivanova K, Marina M, Mitov I, Petrov P, Ozden A, Popova M. The status of antimicrobial resistance of Helicobacter pylori in eastern Europe. Clin Microbiol Infect. 2002 Jul;8(7):388-96. doi: 10.1046/j.1469-0691.2002.00435.x. PMID 12199848